CLINICAL TRIAL: NCT01528059
Title: A Prospective Randomised Study Comparing Billroth II With Roux-en-Y Reconstruction After Radical Distal Subtotal Gastrectomy for Gastric Cancer Comorbid With Type 2 Diabetes
Brief Title: Roux-en-Y Versus Billroth II Reconstruction After Subtotal Gastrectomy in Gastric Cancer Comorbid With Type II Diabetes
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: feng Zheng (Other)
Responsible Party: Sponsor-Investigator, feng Zheng, MD, Xiamen University
Organization: Xiamen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DongFang; FNSP2009Y0039 (Other Grant/Funding Number: Fujian Natural Science Project)
Record Dates: First submitted 2012-02-02; First posted 2012-02-07 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Gastric Cancer; Type 2 Diabetes
Keywords: Diabetes; Gastric cancer; Gastric bypass
MeSH Terms: conditions — Stomach Neoplasms; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Billroth II (Active Comparator): After stomach resection, the remnant stomach is connected to the jejunum.
  Interventions: Procedure: Stomach-small intestine reconstruction
- Roux en Y (Active Comparator): After stomach resection, the remnant stomach is connected to the distal jejunum while duodenum and the proximal jejunum is reconnected to jejunum.
  Interventions: Procedure: Stomach-small intestine reconstruction

INTERVENTIONS:
Procedure: Stomach-small intestine reconstruction — Billroth II or Roux en Y reconstruction will be performed after gastric resection in stomach patients co-morbid with type 2 diabetes

SUMMARY:
Gastric bypass improves glycemic levels in type 2 diabetes. However, the efficacy may be varied by different gastric-small intestine reconstruction used in the procedure. There are reports that Roux en Y reconstruction may give a better result. The purpose of this study is to compare Roux en Y and Billroth II reconstruction in patients with gastric cancer comorbid with type 2 diabetes.

DETAILED DESCRIPTION:
Type 2 diabetes may cause severe complications such as nephropathy and retinopathy. Additionally, it is associated with increased risk for cardiovascular events and diseases. Surgical intervention with gastric bypass has been shown to attenuate glycemic levels in obese patient comorbid with type 2 diabetes. However, since gastric bypass is not a standard procedure, surgical protocol including stomach and small intestine reconstruction may be varied. The investigators and others have found that stomach and small intestine reconstruction may affect the efficacy of diabetic treatment. In this study, the investigators will compare the efficacy of Billroth II and Roux en Y reconstruction on glycemic control in stomach cancer patients with type 2 diabetes. Both Billroth II and Roux en Y are used in stomach-small intestine reconstruction after subtotal gastrectomy. No differences in postoperative outcomes and quality of life have been reported in Billroth II and Roux en Y reconstruction.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Type 2 diabetes
2. Diagnosed with gastric cancer

Exclusion Criteria:

1. Type 1 diabetes
2. Unresectable cancers

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-02 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Glycemic control | 1 year after surgery
  1. Fasting and postprandial glycemic levels, HbA1C
  2. Number of anti-diabetic drugs
  3. Dosage of anti-diabetic drugs

SECONDARY OUTCOMES:
Nutritional status assessment | 1 year after surgery
  1. Body mass index
  2. Anthropometric analysis
  3. Plasma concentrations of albumin, pre-albumin, transferrin,and CRP

CONTACTS AND LOCATIONS:
Overall Officials: Yu Wang, M.D, Principal Investigator — Dongfang Hospital, Xiamen University
Locations (1):
- DongFang Hospital, Fuzhou, Fujian, China